CLINICAL TRIAL: NCT02956759
Title: Early Laser Treatment for Diabetic Eye Disease in China: The PEARL Pilot Randomized Trial
Brief Title: Early Laser Treatment for Diabetic Eye Disease in China : A Pilot Randomized Trial
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Queen's University, Belfast (Other)
Responsible Party: Principal Investigator, Congdon Nathan, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZOC-PEARL STUDY
Record Dates: First submitted 2016-10-12; First posted 2016-11-07 (Estimated); Last update posted 2022-05-09 (Actual); Status verified 2022-03

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; Pan-retinal photocoagulation; proliferative; non-proliferative
MeSH Terms: conditions — Diabetic Retinopathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Early Intervention (Experimental): pan-retinal photocoagulation laser treatment applied to the study eye within 2-4 weeks.
  Interventions: Procedure: Pan-retinal photocoagulation laser treatment
- Standard Care (Active Comparator): pan-retinal photocoagulation laser treatment deferred until the onset of any PDR.
  Interventions: Procedure: Pan-retinal photocoagulation laser treatment

INTERVENTIONS:
Procedure: Pan-retinal photocoagulation laser treatment — PRP initially consists of 1200 - 1600 burns given over 2-3 sessions and separated by2-3weeks by 532-argon laser machine.
  Other Names: PRP laser treatment

SUMMARY:
To compare immediate laser pan-retinal photocoagulation (PRP) treatment of severe or very severe non proliferative diabetic retinopathy (NPDR) stage versus deferral of treatment until the appearance of any proliferative diabetic retinopathy (PDR) in rural and urban patients in China.

Interview data from some patients and survey data from ophthalmologists in the study hospitals will help determine acceptability of early treatment, and how to overcome barriers to increased use of this option.

DETAILED DESCRIPTION:
China now has the world's largest number of diabetic persons. Population studies show that only 10% of Chinese rural-dwellers with DR receive therapy. The current standard approach to treatment of DR often requires patients to return for multiple examinations over years, before they reach trial-proven criteria for treatment. This long process is ill-suited to support good compliance with care in low-resource settings. Our recent published review suggests that earlier PRP treatment, which could reduce the burden of compliance, may be clinically effective and cost effective, but the current evidence base is insufficient to make a firm recommendation.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged >= 18 years with untreated DR at severe or very severe NPDR stage in either one or both eyes, according to the clinical opinion of the investigator.
* Sufficiently clear ocular media to allow visualization of the retina and retinal photography in either eye.
* Capable of giving informed consent.

Exclusion Criteria:

* DR at later stage of retinopathy than severe or very severe (eg, two or more of the 4-2-1 criteria are met) NPDR in either eye, but a patient may be enrolled if one eye has severe or very severe NPDR and the fellow eye has PRP-treated PDR and has been stable after treatment.
* Clinically significant macular edema in either eye.
* Dense cataracts or other media opacity preventing visualization of the retina in the eye.
* History of previous surgical or laser treatment for DR or other retinal conditions in a study eye, including history of anti-VEGF or corticosteroid injection or focal laser for DME within 6 months, or any history of scleral buckle, vitrectomy or other retinal detachment repair.
* History of other retinal vascular disorders including CRVO, CRAO, BRVO, BRAO in the study eye.
* Previous cataract or glaucoma surgery is specifically allowed if performed ≥ 6 weeks prior to enrollment.
* Pregnancy.
* Severe renal insufficiency treated with hemodialysis treatment, kidney transplant, pancreatic transplant, and intensive insulin therapy initiated within 4 months.
* Nystagmus, unable to cooperate with laser treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Proportion of eyes progressing to any degree of PDR | 1 year
  The diagnosis of PDR will be made by detecting either active new vessels in the optic nerve head or elsewhere in the retina as determined by fundus photography read by a masked investigator or preretinal/vitreous haemorrhage at any time during the 12 month follow-up period.

SECONDARY OUTCOMES:
Proportion of early versus standard treated eyes with: Loss of >= 10 and of 15 ETDRS letters | 1 year
Mean change in best corrected visual acuity from baseline to week 52. | 1 year
Proportion of early versus standard treated eyes with: retinal detachment | 1 year
Proportion of early versus standard treated eyes with: increase of diabetic macular edema per Optical Coherence Tomography | 1 year
Sensitivity & specificity of the diagnosis of any degree of PDR among study ophthalmologists | 1 year
  Study ophthalmologists will also ascertain the primary outcome measure (diagnosis of any degree of PDR) on the basis of slit-lamp biomicropscopy fundus examination with a contact lens and indirect ophthalmoscopy. We will compare the sensitivity & specificity of the diagnosis of any degree of PDR among study ophthalmologists with the gold stander (diagnosis provided by graders according to the fundus photos.)

OTHER OUTCOMES:
Comparing the Early versus Standard groups: Proportion of participants show on recommended revisits on time and accept recommended treatments (laser treatment .etc) | 1 year
Patient vision-related quality of life (VRQOL); composite and individual domain scores of the NEI VFQ25 questionnaire. | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Nathan Congdon, PhD, Principal Investigator — Zhongshan Ophthalmic Center, Sun Yat-sen University
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Xu Y, Wang L, He J, Bi Y, Li M, Wang T, Wang L, Jiang Y, Dai M, Lu J, Xu M, Li Y, Hu N, Li J, Mi S, Chen CS, Li G, Mu Y, Zhao J, Kong L, Chen J, Lai S, Wang W, Zhao W, Ning G; 2010 China Noncommunicable Disease Surveillance Group. Prevalence and control of diabetes in Chinese adults. JAMA. 2013 Sep 4;310(9):948-59. doi: 10.1001/jama.2013.168118. PMID 24002281
- [Background] Wang FH, Liang YB, Zhang F, Wang JJ, Wei WB, Tao QS, Sun LP, Friedman DS, Wang NL, Wong TY. Prevalence of diabetic retinopathy in rural China: the Handan Eye Study. Ophthalmology. 2009 Mar;116(3):461-7. doi: 10.1016/j.ophtha.2008.10.003. Epub 2009 Jan 24. PMID 19168222
- [Background] Royle P, Mistry H, Auguste P, Shyangdan D, Freeman K, Lois N, Waugh N. Pan-retinal photocoagulation and other forms of laser treatment and drug therapies for non-proliferative diabetic retinopathy: systematic review and economic evaluation. Health Technol Assess. 2015 Jul;19(51):v-xxviii, 1-247. doi: 10.3310/hta19510. PMID 26173799
- [Background] Shimura M, Yasuda K, Nakazawa T, Kano T, Ohta S, Tamai M. Quantifying alterations of macular thickness before and after panretinal photocoagulation in patients with severe diabetic retinopathy and good vision. Ophthalmology. 2003 Dec;110(12):2386-94. doi: 10.1016/j.ophtha.2003.05.008. PMID 14644723
- [Background] Japanese Society of Ophthalmic Diabetology, Subcommittee on the Study of Diabetic Retinopathy Treatment; Sato Y, Kojimahara N, Kitano S, Kato S, Ando N, Yamaguchi N, Hori S. Multicenter randomized clinical trial of retinal photocoagulation for preproliferative diabetic retinopathy. Jpn J Ophthalmol. 2012 Jan;56(1):52-9. doi: 10.1007/s10384-011-0095-2. Epub 2011 Oct 19. PMID 22009219
- [Background] Fundus photographic risk factors for progression of diabetic retinopathy. ETDRS report number 12. Early Treatment Diabetic Retinopathy Study Research Group. Ophthalmology. 1991 May;98(5 Suppl):823-33. PMID 2062515